CLINICAL TRIAL: NCT05293964
Title: A Multicenter, Open-label, Phase I Clinical Study to Evaluate the Safety, Pharmacokinetics, and Antitumor Efficacy of SIM0270 Alone or in Combination in Subjects with ER-positive, HER-2 Negative Locally Advanced or Metastatic Breast Cancer
Brief Title: Phase I Study to Evaluate SIM0270 Alone or in Combination in ER+, HER2- Locally Advanced or Metastatic Breast Cancer
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Jiangsu Simcere Pharmaceutical Co., Ltd. (Industry)
Collaborators: Nanjing Zaiming Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: SIM-1907-02-SERD-101
Record Dates: First submitted 2022-03-07; First posted 2022-03-24 (Actual); Last update posted 2024-11-29 (Actual); Status verified 2024-11

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — palbociclib; Everolimus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- SIM0270 (Experimental): Phase Ia SIM0270 monotherapy dose escalation and expansion
  Interventions: Drug: SIM0270
- SIM0270+palbociclib (Experimental): Phase Ib SIM0270 with palbociclib dose escalation and expansion
  Interventions: Drug: SIM0270; Drug: Palbociclib
- SIM0270+everolimus (Experimental): Phase Ib SIM0270 with everolimus dose escalation and expansion
  Interventions: Drug: SIM0270; Drug: everolimus

INTERVENTIONS:
Drug: SIM0270 — SIM0270 is an oral, selective estrogen receptor degrader (SERD)
  Other Names: SCR6852
Drug: Palbociclib — palbociclib is a selective inhibitor of cyclin D-cyclin-dependent kinase (CDK) 4/6
  Arms: SIM0270+palbociclib
Drug: everolimus — Everolimus is an inhibitor of mTOR (mammalian target of rapamycin)
  Arms: SIM0270+everolimus

SUMMARY:
This study is a multi-center, open-label, Phase 1 clinical study to evaluate the safety, pharmacokinetic (PK) and anti-tumor efficacy of SIM0270 and SIM0270 in combination with palbociclib or everolimus in subjects with estrogen receptor (ER) -positive, human epidermal growth factor receptor (HER-2) -negative locally advanced or metastatic breast cancer.

DETAILED DESCRIPTION:
The study is comprised of two parts: Phase Ia and Phase Ib. Phase Ia includes dose-escalating stage and dose expansion stageof SIM0270 monotherapy to determine the MTD/ RP2D and the preliminary safety and efficacy of SIM0270; Phase Ib includes 2 arms, armA: dose escalation and dose expansion of SIM0270 in combination with palbociclib; armB: dose escalation and dose expansion of SIM0270 in combination with palbociclib everolimus; phase Ib is designed to determine the MTD/RP2D and the preliminary safety and efficacy of SIM0270 in combination with palbociclib or everolimus.

ELIGIBILITY:
key Inclusion Criteria:

1. voluntary participation in clinical trials and signature of informed consent.
2. age ≥ 18 years, male or female.
3. Histologically or cytologically confirmed metastatic/locally advanced ER-positive, HER-2 negative breast cancer subjects.
4. previous treatment meets the criteria of the protocol defined.
5. ECOG score of 0 or 1 .
6. at least one measurable lesion that meets RECISTv1.1 criteria. Osteolytic lesions can be included in the Ia dose-escalating .
7. expected survival ≥ 12 weeks.
8. Adequate organ and bone marrow function.
9. Women of childbearing potential must have a negative serum pregnancy test within 7 days prior to the first dose.
10. Postmenopausal women; Premenopausal or perimenopausal female subjects met protocol requirements.

key Exclusion Criteria:

1. Documented medical history or ongoing gastrointestinal disease or other malabsorption that may affect the absorption of oral study drug.
2. Participated in other clinical trials of investigational drugs or investigational devices within 28 days before the first medication; or received chemotherapy, targeted therapy, immunotherapy and clinical trial medication and other anti-tumor treatment within 4 days or 5 half-lives of the first medication (whichever is shorter), or received radiotherapy, endocrine drugs or Chinese patent medicines with anti-tumor indications 2 weeks before the first medication;
3. The toxicity of previous anti-tumor treatment has not recovered to grade 0 or 1 (alopecia, chemotherapy-induced peripheral neurotoxicity ≤ grade 2 can be included).
4. Major surgical surgery (except biopsy) or incomplete healing of the surgical incision 4 times before the first study drug treatment;
5. Known other malignant tumors within 2 years before enrollment (except treated basal cell carcinoma, scaly cell carcinoma and/or radical carcinoma in situ);
6. Leptomeningeal metastasis confirmed by MRI or known cytology of CSF, or cranial Increased internal pressure or brain metastases with unstable central nervous symptoms (within 2 weeks prior to initial medication Treatment with any craniotropic, glucocorticokinin, or anticonvulsant);
7. Previous history of interstitial lung disease, drug-induced interstitial lung disease, symptomatic interstitial lung disease or any evidence of active pneumonia on chest CT scan 4 before the first study drug treatment;
8. known to interfere with the test requirements of mental illness or drug abuse disease.
9. History of human immunodeficiency virus HIV infection, or active bacterial or fungal infection requiring systemic treatment .
10. presence of active syphilis infection.
11. Subjects with known active hepatitis B virus (HBV) or hepatitis C virus (HCV) infection with abnormal liver function.
12. History of clinically significant cardiovascular disease.
13. History of serious allergic reactions to the study drugs or excipients used in the protocol.
14. Women who are pregnant or lactating.
15. Prior use of SERD oral medications.
16. Subjects who use drugs or herbal supplements known to be moderate/strong inhibitors of CYP3A 2 Weeks before the first dose.Or Subjects who use drugs or herbal supplements known to be moderate/strong inducers of CYP3A 4 weeks before the first dose.
17. Other conditions that the investigator considers unsuitable for this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 214 (Actual)
Dates: Start 2022-05-18 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2025-09-08 (Estimated)

PRIMARY OUTCOMES:
Maximum Tolerated Dose | At the end of Cycle 1 (each cycle is 28 days)
  Dose Escalation: Maximum Tolerated Dose (MTD) of SIM0270 When Administered as a Single Agent or in Combination with Palbociclib or Everolimus
recommended phase 2 Dose | At the end of Cycle 1 (each cycle is 28 days)
  Dose Escalation: recommended phase 2 Dose (RP2D) of SIM0270 When Administered as a Single Agent or in Combination with Palbociclib or Everolimus
Dose-Limiting Toxicities | At the end of Cycle 1 (each cycle is 28 days)
  Dose Escalation: Number of Participants with Dose-Limiting Toxicities When SIM0270 is Administered as a Single Agent or in Combination with Palbociclib or Everolimus

SECONDARY OUTCOMES:
Adverse event | From Baseline until 30 days after the last dose of study treatment
  Number of Participants with Adverse Events by Severity, According to National Cancer Institute Common Terminology Criteria for Adverse Events version 5.0 (NCI-CTCAE v5.0)
Peak Plasma Concentration (Cmax) of SIM0270 as monotherapy or combination with palbociclib or everolimus | At the end of Cycle 4 (each cycle is 28 days)
  Peak Plasma Concentration (Cmax)
Time of Peak Plasma Concentration (Tmax) of SIM0270 as monotherapy or combination with palbociclib or everolimus | At the end of Cycle 4 (each cycle is 28 days)
  Time of Peak Plasma Concentration (Tmax)
Area under the plasma concentration versus time curve (AUC) of SIM0270 as monotherapy or combination with palbociclib or everolimus | At the end of Cycle 4 (each cycle is 28 days)
  Area under the plasma concentration versus time curve (AUC)
clinical benefit rate | through study completion, an average of 1 year
  Antitumour activity by evaluation of clinical benefit rate assessments using Response Evaluation Criteria in breast cancer (RECIST 1.1)or Response Assessment in Neuro-Oncology Brain Metastases (RANO-BM)
disease control rate | through study completion, an average of 1 year
  Antitumour activity by evaluation of disease control rate assessments using Response Evaluation Criteria in breast cancer (RECIST 1.1)or Response Assessment in Neuro-Oncology Brain Metastases (RANO-BM)
duration of response | through study completion, an average of 1 year
  Antitumour activity by evaluation of duration of response assessments using Response Evaluation Criteria in breast cancer (RECIST 1.1)or Response Assessment in Neuro-Oncology Brain Metastases (RANO-BM)
progression free survival | From date of C1D1 until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 100 months
  Antitumour activity by evaluation of progression free survival assessments using Response Evaluation Criteria in breast cancer (RECIST 1.1)or Response Assessment in Neuro-Oncology Brain Metastases (RANO-BM)
time to progression | From date of C1D1 until the date of first documented progression, assessed up to100 months
  Antitumour activity by evaluation of time to progression assessments using Response Evaluation Criteria in breast cancer (RECIST 1.1)or Response Assessment in Neuro-Oncology Brain Metastases (RANO-BM)
time to response | through study completion, an average of 1 year
  Antitumour activity by evaluation of time to response assessments using Response Evaluation Criteria in breast cancer (RECIST 1.1)or Response Assessment in Neuro-Oncology Brain Metastases (RANO-BM)
overall survival | From date of C1D1 until the date of death from any cause, assessed up to 100 months
  Antitumour activity by evaluation of overall survival assessments
overall response rate | through study completion, an average of 1 year
  Antitumour activity by evaluation of tumour response assessments using Response Evaluation Criteria in breast cancer (RECIST 1.1)

CONTACTS AND LOCATIONS:
Overall Officials: Jiong Wu, phD, Principal Investigator — chief physician
Locations (1):
- Fudan University Shanghai Cancer Center, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No
the plan to make individual participant data (IPD) available to other researchers is not decided yet.